CLINICAL TRIAL: NCT03474562
Title: Effect of High-Dose Rosuvastatin Combined With Telmisartan or Amlodipine on Glucose Metabolism in Atherosclerotic Cardiovascular Disease (ASCVD) Patients With Impaired Fasting Glucose (IFG) and Hypertension: A Randomized, Open-Label, Parallel, Prospective Study
Brief Title: High-Dose Statin Combined With Telmisartan vs Amlodipine on Glucose Metabolism in ASCVD Patients With IFG and Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC032
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: ASCVD; Impaired Fasting Glucose; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duowell Tab (Experimental): Telmisartan 40mg/Rosuvastatin 20mg qd for 24 weeks
  Interventions: Drug: Duowell®
- Monorova Tab + Amlopin Tab (Active Comparator): Rosuvastatin 20mg + Amlodipine 5mg qd for 24 weeks
  Interventions: Drug: Monorova® + Amlopin®

INTERVENTIONS:
Drug: Duowell® — Telmisartan/Rosuvastatin 40/20mg (increased to Telmisartan 80mg if SBP > 140mmHg or DBP > 90mmHg at week 12)
  Arms: Duowell Tab
Drug: Monorova® + Amlopin® — Rosuvastatin 20mg + Amlodipine 5mg (increased to Amlodipine 10mg if SBP > 140mmHg or DBP > 90mmHg at week 12)
  Arms: Monorova Tab + Amlopin Tab

SUMMARY:
This study will evaluate the effect of high-dose rosuvastatin combined with telmisartan or amlodipine on glucose metabolism in ASCVD patients with impaired fasting glucose and hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged 19 to 75 years
3. Patients with ASCVD requiring high-intensity statin therapy (in accordance with the clinical ASCVD diagnostic criteria in the 2013 ACC/AHA Guideline)

   - Coronary artery disease
   * acute coronary syndrome
   * history of myocardial infarction (MI)
   * stable or unstable angina
   * history of coronary revascularization
   * stroke or transient ischemic attack (TIA)
   * peripheral arterial disease, history of peripheral arterial revascularization
4. Those who are taking antihypertensive drugs, or SBP > 140mmHg or DBP > 90mmHg on the left side
5. High-risk group (except for gestational diabetes) who has not been diagnosed with diabetes before, and who falls under one of the following criteria:

   * impaired fasting glucose (IFG): 100-125 mg/dL (5.6-6.9 mmol/L)
   * impaired glucose tolerance (IGT): plasma blood glucose 140-199mg/dL (7.8 to 11.0 mmol/L) 2 hours after oral administration of glucose 75g
   * HbA1c: 5.7-6.4%

Exclusion Criteria:

1. Those who are treated with secondary hypertension or malignant hypertension
2. Uncontrollable diabetes with HbA1c ≥ 10%
3. Total cholesterol ≥ 300mg/dL
4. Fasting LDL-C ≤ 70 mg/dL
5. Fasting triglyceride ≥ 500 mg/dL
6. History of muscular disease or rhabdomyolysis due to use of statin
7. Hypersensitive to statin or ARBs
8. Contraindications stated in the SPC of telmisartan or rosuvastatin including the following:

   * severe renal disease (CrCL < 30mL/min: Cockcroft-gault formula or estimated GFR (MDRD) < 30mL/min/1.73m2)
   * ALT, AST > 3x ULN or history of active liver disease
   * CPK > 3x ULN
   * hyperkalemia with serum K > 5.5 mEq/l
9. Those who are participating in clinical trials of other investigational products
10. Those who cannot discontinue all other treatment for hypertension or hyperlipidemia than the investigational products, and concomitant medications and supplements that can affect the therapeutic effect of hypertension and hyperlipidemia during the trial period
11. Other than the above who is deemed to be ineligible to participate in the trial by investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in homeostasis model assessment for insulin resistance (HOMA-IR) | Baseline, Week 24

SECONDARY OUTCOMES:
Change from baseline to week 12 and week 24 in HOMA-IR | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in fasting plasma glucose (FPG) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in insulin level | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in homeostatic model assessment for β-cell function (HOMA-B) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in hemoglobin A1c (HbA1c) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), and low-density lipoprotein cholesterol (LDL-C) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in C-reactive protein (CRP) | Baseline, Week 12, Week 24

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Dankook University Hospital, Cheonan
  - Gangnam Severance Hospital, Seoul
  - Severance Hospital, Seoul